CLINICAL TRIAL: NCT01937572
Title: Visionaire Versus Conventional Knee Arthroplasty: A Prospective Study
Brief Title: Visionaire: A Prospective Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: An interim analysis found the study would not be able to reach significance without a large increase in subjects which was not feasible.
Sponsor: The Hawkins Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Pro00013735
Record Dates: First submitted 2013-08-28; First posted 2013-09-09 (Estimated); Last update posted 2018-07-05 (Actual); Status verified 2018-07

CONDITIONS: Osteoarthritis
Keywords: Total knee arthroplasty (TKA); Computer aided systems
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Computer-aided TKA (Experimental): The Visionaire system is a computer-aided system utilizing MRI of the knee prior to TKA surgeries. This technology achieves accurate rotational and A-P position. All of the commonly-referred anatomical landmarks (AP axis, epicondylar axis) are analyzed pre-operatively, allowing for the proper positioning of the implant for each patient.
  Interventions: Other: Visionaire system (Knee MRI)
- Conventional TKA (Other): A conventional TKA utilizes a jig system based on either intra-medullary or extra-medullary guides. No knee MRI is utilized for a conventional TKA.
  Interventions: Other: No Knee MRI

INTERVENTIONS:
Other: Visionaire system (Knee MRI)
  Other Names: Visionaire
  Arms: Computer-aided TKA
Other: No Knee MRI
  Arms: Conventional TKA

SUMMARY:
The purpose of the current study is to validate the technology of MRI-based alignment for total knee replacements and to collect data on potential advantages of the computer aided system.

1. It is hypothesized that there will be no significant differences in position, loosening, or function of the Visionaire total knee as compared to the conventional total knee.
2. It is hypothesized that the Visionaire total knee will be significantly better with regard to operative time, tourniquet time, blood loss, and procedural set-up, turnover time, and overall costs.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with sufficient symptoms from articular knee pathology to be an appropriate candidate for TKA

Exclusion Criteria:

* prior TKA
* ipsilateral upper tibial or distal femoral osteotomy
* ipsilateral total hip arthroplasty
* patient with significant >15o varus or valgus
* morbid obesity or those patients unable to have an MRI based on thigh circumference (22 cm or less)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2011-11; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Knee Society Score | one year

SECONDARY OUTCOMES:
Degrees off normal AP and lateral alignment | one year

OTHER OUTCOMES:
Total blood loss | two days
Operative time | one day
Operative room setup and turnover times | one day
Procedural cost | one day

CONTACTS AND LOCATIONS:
Overall Officials: Brian Burnikel, MD, Principal Investigator — Steadman Hawkins Clinic of the Carolinas - Greenville Hospital System
Locations (1):
- Steadman Hawkins Clinic of the Carolinas - Greenville Hospital System, Greenville, South Carolina, United States